CLINICAL TRIAL: NCT04940663
Title: Neurobehavioral Mechanisms of Social Isolation and Loneliness in Serious Mental Illness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Daphne Holt, Associate Professor of Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021P001826
Record Dates: First submitted 2021-06-18; First posted 2021-06-25 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Psychosis; Schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ecological Momentary Assessment (Other): EMA collected daily (4x/day) for two weeks
  Interventions: Behavioral: EMA

INTERVENTIONS:
Behavioral: EMA — Participants will complete surveys about their feelings and social habits through a smartphone app (EMA)

SUMMARY:
The proposed research will test the hypothesis that objective social isolation and loneliness are linked to neurobehavioral mechanisms involved in social perception and motivation in individuals with and without serious mental illness. Moreover, it will investigate the specific dynamic interactions among these experiences in daily life and how they, and their neurobehavioral predictors, are linked to day-to-day functioning. The findings of this project could provide novel targets for therapeutics aimed at improving functioning and overall quality of life in individuals with serious mental illnesses, as well as quantitative phenotypes for use in early detection efforts.

DETAILED DESCRIPTION:
Some of the most debilitating and harmful aspects of serious mental illnesses (SMI) are the 1) social isolation (low numbers of social contacts) and 2) the subjective experiences of social disconnection (loneliness) that frequently accompany these conditions. Social isolation and loneliness greatly impact day-to-day functioning and are associated with poor cardiometabolic health and early mortality in SMI, and currently there are no available treatments that can prevent or reverse these devastating consequences of having these illnesses. This may be in part because the neural and psychological mechanisms underlying social isolation and loneliness in SMI, and how they impact functioning and health outcomes, are poorly understood. However, recent clues from studies employing advanced neuroimaging and digital assessments have formed the basis of a novel approach to investigating such mechanisms, outlined in this proposal. Prior work has indicated that objective isolation and loneliness are correlated but also somewhat independent. Recent neuroimaging findings support this model, revealing that social isolation and loneliness have both shared and distinct neural correlates. However, it is also clear that these are not static phenomena; smartphone-based assessments have revealed transient, dynamic changes in social isolation and loneliness. Individual differences in the anticipation of rejection are associated with momentary experiences of loneliness, greater avoidance and subsequent increases in social isolation. Thus, in the current application, we propose to comprehensively measure both the relatively stable neural and behavioral predictors of social isolation and loneliness, as well as the moment-to-moment changes in these experiences, in 60 individuals with SMI and 60 control subjects. In Aim 1 of the proposed project, we will show that the higher levels of social isolation and loneliness in SMI are linked to shared and distinct neural responses to social stimuli, with deficient responses of social perception-related circuitry (medial temporal lobe regions) linked to social isolation, and deficient responses of reward-related circuitry (basal ganglia regions) linked to loneliness. In Aim 2, we will measure transient changes in social isolation and loneliness with smartphone assessments using a longitudinal "burst" design. Lastly, in Aim 3, we will determine how the quantitative markers of social isolation and loneliness identified in Aims 1 and 2 predict indices of real-world functioning, measuring the stability of these associations over time. Thus, in this project, we will show that fundamental neural and behavioral processes drive momentary variation in the experience of social isolation and loneliness, and directly impact functioning in SMI. In follow-up work, these findings can be used as objective targets in studies of novel interventions which aim to address these major causes of disability.

ELIGIBILITY:
Inclusion Criteria:

1. 18-55 years old
2. Experienced a psychotic disorder or mood disorder

Exclusion Criteria:

1. Any neurological disorder or current substance use disorder (during the past 6 months)
2. Not proficient in English
3. A recent change in medication, or an acute symptom presentation
4. Standard exclusion criteria for participation in an MRI scan (e.g., presence of metal in the body, claustrophobia, a history of head trauma).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Trait level social isolation and loneliness | 6 months
  UCLA Loneliness Scale(20 and 4 item), Social Network Index, Social Anhedonia Scale, Penn facial affect recognition Task, Social Disconnectedness Scale, Social Provisions Scale
Characterize within-person, dynamic changes in objective isolation and loneliness | 6 months
  EMA questions derived from the UCLA Loneliness Scales, perceived discrimination scale
Psychosocial functioning | 6 months
  Quality of Life Scale, Cornblatt Global Functioning - Social and Role Scales
Physical health and cardiometabolic/immunological panel | 6 months
  Height, weight, waist circumference, systolic and diastolic blood pressure, blood oxygen level, heart rate, interleukin-6, TNF-alpha, Complete metabolic panel, lipid panel, C-reactive protein, Cortisol, CBC, HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Daphne J Holt, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States